CLINICAL TRIAL: NCT06678321
Title: THE EFFECT OF THE MOBILE GAME "ASK OLSUN!" ON THE DEVELOPMENT OF YOUNG ADULTS' ATTITUDES AND PERCEPTIONS TOWARDS DATING VIOLENCE: A RANDOMIZED CONTROLLED STUDY"
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Funda Yıldız, Lecturer, Eskisehir Osmangazi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: FUNDAYILDIZ
Record Dates: First submitted 2024-11-06; First posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Dating Violence
Keywords: dating violence; mobil game; university students

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- İntervention group (Experimental): Mobil Game
  Interventions: Behavioral: Mobil game
- Control group (No Intervention): No game

INTERVENTIONS:
Behavioral: Mobil game — Participants in the intervention group will be asked to play the game and complete all parts.
  Arms: İntervention group

SUMMARY:
This research; It was designed as a 3-stage study with the aim of evaluating the mobile game that will be developed to positively change the attitudes and perceptions of young people studying at Istanbul Bilgi University towards dating violence. The first phase of the research was designed in a cross-sectional pattern to determine young people's general attitudes towards dating violence and their perceptions towards dating violence. The second phase of the study was designed in a methodological pattern to include the development of a mobile game to positively change young people's general attitudes and perceptions towards dating violence and increase their awareness. The third phase of the study was designed with a randomized controlled experimental design to determine the effect of the developed mobile game on young people's general attitudes towards dating violence and their perceptions towards dating violence. In the study, "Socio-demographic Characteristics and Data Form" created by the researcher will be used to collect data, "Flirting Violence Attitude Scale" will be used to determine the general attitude towards dating violence, and "Flirting Violence Perception Scale" will be used to determine the perception of dating violence. "Socio-demographic Data Form", Dating Violence Attitude Scale and Dating Violence Perception Scale will be used in the second stage of the study to recruit participants to the study groups. Research data will be collected online by the researcher via Google surveys after the participants are informed about the research and their consent is obtained.

In the third stage of the study, data will be collected in two separate processes: pre-test and post-test. The pre-test consists of the Sociodemographic Characteristics and Data Form, the Dating Violence Attitude Scale and the Dating Violence Perception Scale. The pre-test will be administered after oral and written consent of the participants included in the intervention and control groups is obtained.

In the last test; The Dating Violence Attitude Scale and the Dating Violence Perception Scale will be used. The post-test will be administered after oral and written consent of the participants included in the study groups is obtained.

A mobile game consisting of 8 episodes within the scope of dating violence based on the health belief model will be played to the intervention group and the final test will be applied to the same group 4 weeks later. There will be no intervention in the control group, and the final test will be administered 4 weeks later.

DETAILED DESCRIPTION:
This research; It was designed as a 3-stage study with the aim of evaluating the mobile game that will be developed to positively change the attitudes and perceptions of young people studying at Istanbul Bilgi University towards dating violence. The first phase of the research was designed in a cross-sectional pattern to determine young people's general attitudes towards dating violence and their perceptions towards dating violence. The second phase of the study was designed in a methodological pattern to include the development of a mobile game to positively change young people's general attitudes and perceptions towards dating violence and increase their awareness. The third phase of the study was designed with a randomized controlled experimental design to determine the effect of the developed mobile game on young people's general attitudes towards dating violence and their perceptions towards dating violence. In the study, "Socio-demographic Characteristics and Data Form" created by the researcher will be used to collect data, "Flirting Violence Attitude Scale" will be used to determine the general attitude towards dating violence, and "Flirting Violence Perception Scale" will be used to determine the perception of dating violence. "Socio-demographic Data Form", Dating Violence Attitude Scale and Dating Violence Perception Scale will be used in the second stage of the study to recruit participants to the study groups. Research data will be collected online by the researcher via Google surveys after the participants are informed about the research and their consent is obtained.

In the third stage of the study, data will be collected in two separate processes: pre-test and post-test. The pre-test consists of the Sociodemographic Characteristics and Data Form, the Dating Violence Attitude Scale and the Dating Violence Perception Scale. The pre-test will be administered after oral and written consent of the participants included in the intervention and control groups is obtained.

In the last test; The Dating Violence Attitude Scale and the Dating Violence Perception Scale will be used. The post-test will be administered after oral and written consent of the participants included in the study groups is obtained.

A mobile game consisting of 8 episodes within the scope of dating violence based on the health belief model will be played to the intervention group and the final test will be applied to the same group 4 weeks later. There will be no intervention in the control group, and the final test will be administered 4 weeks later.

ELIGIBILITY:
Inclusion Criteria:

* Having at least one dating relationship
* Being exposed to dating violence (any type) at least once in a dating relationship
* Be single

Exclusion Criteria:

* Married
* Have never been in a dating relationship
* Not having experienced dating violence in any way
* Not volunteering to participate in the research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2024-11-20 (Estimated); Primary Completion 2025-06-20 (Estimated); Study Completion 2025-06-20 (Estimated)

PRIMARY OUTCOMES:
Dating Violence Perception Scale (DVPS) | Baseline and after 4 weeks
  The scale consists of 3 sub-dimensions including items related to physical, sexual and psychological dating violence and 15 items in each sub-dimension. The score that can be obtained from the scale varies between 15 and 90. There are 3 reverse items in the scale. The high score obtained from the scale shows that the person cares about dating violence and does not perceive it as a big problem.
Dating Violence Attitude Scale (DVAS) | Baseline and after 4 weeks
  The scale includes physical, emotional, economic, sexual and general violence sub-dimensions.
  It is a 5-point Likert-type scale scored between 1-5 and consists of 28 items (1: Strongly disagree, 2: Disagree, 3: Undecided, 4: Agree, 5: Strongly agree).
  When the scores obtained from the scale approach 1, it indicates that the individual has an attitude in favour of dating abuse.

CONTACTS AND LOCATIONS:
Locations (1):
- Funda Yıldız, Şişli, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://cinselsiddetlemucadele.org/ne-var-ne-yok-genclik-calismalari/